CLINICAL TRIAL: NCT04572568
Title: Registry of Multimodality Treatment for Brain Arteriovenous Malformation in Mainland China
Acronym: MATCH
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Neurosurgical Institute (Other); Peking University International Hospital (Other); West China Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Sichuan Provincial People's Hospital (Other); The First Hospital of Jilin University (Other); Shanxi Provincial People's Hospital (Other Government); The Second Hospital of Shandong University (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The General Hospital of Central Theater Command (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Tianjin Medical University Second Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Shengjing Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Hainan People's Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Second Xiangya Hospital of Central South University (Other); Second Affiliated Hospital of Soochow University (Other); General Hospital of Ningxia Medical University (Other); Lanzhou University Second Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); Qilu Hospital of Shandong University (Other); Jining Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Shandong Provincial Hospital (Other Government); The Affiliated Hospital of Xuzhou Medical University (Other); Henan Provincial People's Hospital (Other); Binzhou Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: KY 2020-003-01
Record Dates: First submitted 2020-09-07; First posted 2020-10-01 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Brain Arteriovenous Malformation
Keywords: Brain Arteriovenous Malformation; multi-disciplinary treatment; embolization; stereotactic radiosurgery; microsurgical resection; hybrid surgery; conservative/medical treatment; hemodynamic; outcomes; subsequent hemorrhage; obliteration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: Ruptured AVMs:
  1. AVMs not involved vital eloquent areas, or more than 5 mm away from functional fiber bundles, microsurgery or hybrid surgery can be performed;
  2. Targeted embolization for hemorrhagic predictors could be considered as a monotherapy; embolization can be used as an adjunctive strategy to reduce flow or volume before microsurgery or stereotactic radiosurgery (SRS).
  3. SRS for patients with a volume less than 10ml and not in the acute phase(< 3months) of hemorrhage. Volume-stage or dose-stage can be used for giant AVMs involving important eloquent areas.
  4. Conservation can be used for AVMs that are prone to severe disability due to intervention.
  Unruptured AVMs:
  Interventions are recommended if unruptured AVMs are assessed as being at high rupture risk, or have refractory epilepsy or acceptable postoperative neurological deficits, otherwise conservative treatment is recommended. The choice of intervention strategy was the same as for ruptured AVM.
  Interventions: Other: Multi-disciplinary assessment
- control group: Patients who had not received a multidisciplinary assessment to develop a treatment plan were included in the control group. It should be noted that the multidisciplinary team for AVM was formed in June 2018, so the prospective AVM cohort from August 2011 to June 2018 and the AVM cohort after June 2018 without comprehensive evaluation of treatment regimens by the multidisciplinary team served as the control group.

INTERVENTIONS:
Other: Multi-disciplinary assessment — 1. Comprehensive evaluation by multidisciplinary experts;
  2. Preoperative multi-modal imaging examination was applied to determine the angioarchitecture, functional fiber bundle, and hemodynamics.
  Groups: experimental group

SUMMARY:
This study is a multi-center, prospective, registry study. This research was supported by the National Key Research and Development Program. They were divided into experimental group and control group according to whether the treatment plan was formulated by a multidisciplinary team. Patients of experimental group is strictly in accordance with standardized multi-disciplinary treatment protocols and meet the following criteria: 1. A multi-disciplinary conference discussion; 2. Detailed preoperative evaluation based on CT, MRI, fMRI and DSA. 3. Treatment modalities meet the following treatment criteria（craniotomy, embolization and stereotactic radiosurgery）. The control group was patients who had not been treated according to a multi-disciplinary treatment protocol.

Patient baseline data, AVM angioarchitectural features, imaging DICOM data, surgical information, and follow-up information were registered. All patients were evaluated for neurofunction at baseline, 3 months, 12 months, and 3 years after treatment. Main observation endpoints: 1. Modified Rankin Scale; 2. Obliteration rate; 3. Subsequent hemorrhage; 4. Complication rate (such as morbidity rate, new-onset neurological dysfunction, and radiation-related complications). Secondary observation endpoint: improvement of clinical symptoms (epilepsy, headache, neurological dysfunction) at 3 months, 12 months, and 3 years after treatment.

DETAILED DESCRIPTION:
This study is a multi-center, prospective registry study led by Beijing Tiantan Hospital, and a number of comprehensive hospitals in mainland China, aiming to uncover the long-term outcomes of AVM in Real-World in China and to discover a standardized diagnosis and treatment process for the comprehensive treatment of brain AVMs. This study is an observational study that will last for 20 years. All patients were enrolled prospectively, and the study will not influence the choice of treatment modalities.

The study cohort of this study was AVM patients aged 1-80 years. The inclusion criteria were as follows: 1. The diagnosis of AVM was confirmed with digital subtraction angiography (DSA) and/or magnetic resonance imaging(MRI); 2.Patients with complete clinical and imaging data; 3. Patient or patient's legal representative agreed to collection of information for this study and signed informed consent. The exclusion criteria were as follows: 1. Received other treatment (surgery, embolization or SRS)before inclusion; 2. Expected survival time is less than 6 months; 3. Spinal AVMs; 4. Patients missing critical baseline and imaging data.

Patients will be divided into two groups: experimental group and control group. Experimental group: Patients who had received a multidisciplinary assessment to develop a treatment plan were included in the experimental group. The details were as follows: Ruptured AVMs: 1. AVMs not involved vital eloquent areas, or more than 5 mm away from functional fiber bundles, microsurgery or hybrid surgery can be performed; 2. Targeted embolization for hemorrhagic predictors could be considered as a monotherapy; embolization can be used as an adjunctive strategy to reduce flow or volume before microsurgery or stereotactic radiosurgery (SRS); 3. SRS for patients with a volume less than 10ml and not in the acute phase(< 3months) of hemorrhage. Volume-stage or dose-stage can be used for giant AVMs involving important eloquent areas; 4.Conservation can be used for AVMs that are prone to severe disability due to intervention. Unruptured AVMs: Interventions are recommended if unruptured AVMs are assessed as being at high rupture risk, or have refractory epilepsy or acceptable postoperative neurological deficits, otherwise conservative treatment is recommended. The choice of intervention strategy was the same as for ruptured AVM. Control group: Patients who had not received a multidisciplinary assessment to develop a treatment plan were included in the control group. It should be noted that the multidisciplinary team for AVM was formed in June 2018, so the prospective AVM cohort from August 2011 to June 2018 and the AVM cohort after June 2018 without comprehensive evaluation of treatment regimens by the multidisciplinary team served as the control group.

An electronic data capture system (EDC) was developed and used for data collection. All the clinical baseline data and imaging data were stored through a cloud server to facilitate the input work at different locations and at different times. Follow-up was conducted at the first 3-6 months and annually after surgery by clinical visit and telephone interview. The evaluation of mRS score was conducted by neurosurgeons who have at least 5 years' experience of clinical practice and all the images were interpreted by at least 2 radiologists independently who are with at least 5 years of clinical experience in radiology center of our institute. Researchers who performed follow-up assessments were blinded to treatment modalities.

The primary outcomes were as follows: modified Rankin Scale, obliteration rate, subsequent hemorrhage, complication rate (such as morbidity rate, new-onset neurological dysfunction, and radiation-related complications) at 3 months, 12 months, and 3 years after treatment. The secondary outcomes were as follows: improvement of clinical symptoms (epilepsy, headache, neurological dysfunction) at 3 months, 12 months, and 3 years after treatment.

Through the final follow-up data, we could compare the short-term outcomes and long-term outcomes between experimental and control group. In addition, intra-group comparisons can be made among subgroups of different intervention strategies to explore the best individualized treatment strategies for different AVM patients.

Treatment criteria for craniotomy: 1. For patients with a history of rupture and bleeding: a. If the lesion is not located in the deep functional area, surgical treatment is recommended; b. If the lesion is multi-system blood supply or high blood flow, the volume is large, and with a deep blood supply, hybrid surgery (embolization + resection) can be performed; c. If the lesion is located in the deep functional area, craniotomy is not recommended. 2. For patients with unruptured hemorrhage: a. If the lesion is not located in the deep brain tissue, and is not located in an important functional area or the fiber bundle is more than 5mm away from the lesion, then surgery or combined surgery can be performed; b. If the lesion is located in the deep brain tissue, important functional areas or fiber bundles are less than 5mm away from the lesion, craniotomy is not recommended; c. If the lesion does not have the above characteristics, surgical resection alone can be performed.

Interventional embolization treatment standards: 1. Ruptured bAVM should be actively treated. If there is no need for craniotomy to clear the hematoma in the acute phase, DSA should be performed 2-6 weeks after hemorrhage, and individualized treatment plans should be developed and actively treated. 2. Unruptured bAVM, if there are bleeding-related risk factors (aneurysm or high-flow fistula), relevant risk factors should be actively treated; When stereotactic radiation is planned, when craniotomy or SRS was planned, preoperative embolization for flow reduction or volume reduction is recommended; 3. Unruptured bAVM, without the above risk factors, conservative treatment was suggested if symptoms could be well controlled.

Stereotactic radiosurgery standard treatment: 1. No history of bleeding: Patients with no indications for craniotomy and with appropriate volume for radiosurgery, and poor symptom controlled. Pre-treatment imaging assessment DSA (required) and enhanced MRI was required to clarify the structure of the malformation; 2. There is a history of bleeding: the period between bleeding time and the time of consultation is less than 3 months, it is recommended to wait head-enhanced MRI and DSA were performed after the hemorrhage was absorbed (3 months) to confirm the vascular architecture. 3.Volume-stage or dose-stage can be used for giant AVMs involving important eloquent areas.

Conservation standard treatment: 1. Ruptured AVMs: Patients prone to severe disability due to intervention; 2. Unruptured AVMs: Patients were assessed as having a low rupture risk, or without refractory epilepsy or with a high risk of postoperative neurological deficits.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of AVM was confirmed with digital subtraction angiography (DSA) and/or magnetic resonance imaging(MRI).
2. Patients with complete clinical and imaging data.
3. Patient or patient's legal representative agreed to collection of information for this study and signed informed consent.

Exclusion Criteria:

1. Received other treatment (surgery, embolization or SRS)before inclusion;
2. Expected survival time is less than 6 months;
3. Spinal AVMs;
4. Patients missing critical baseline and imaging data.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the diagnosis of AVM was confirmed with digital subtraction angiography (DSA) and/or magnetic resonance imaging(MRI).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-08-01 (Actual); Primary Completion 2032-04-01 (Estimated); Study Completion 2033-04-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 3 months, 1 year, and 3 years after treatment
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
obliteration rate | 3 months, 1 year, and 3 years after treatment
  Complete obliteration of the nidus was confirmed by DSA or MRA, then compare the obliteration rate between each group.
subsequent hemorrhage | 3 months, 1 year, and 3 years after treatment
  Intracranial hemorrhage that could be attributed to AVMs, and can be confirmed by CT and other imaging.
complication rate | 3 months, 1 year, and 3 years after treatment
  such as morbidity rate, new-onset neurological dysfunction, and radiation-related complications

SECONDARY OUTCOMES:
Improvement of epilepsy | 3 months, 1 year, and 3 years after treatment
  Improvement of epilepsy at 3 months, 1 year, and 3 years after treatment The prognosis of epilepsy was assessed by Engle classification: Grade I, the seizures disappear completely or only with aura; Grade II, the seizures are very few (≤3 times/year); Grade III, the seizures are >3 times/year, but the seizures are reduced by ≥75%; Grade IV, the seizures are reduced <75 %.
Improvement of headache | 3 months, 1 year, and 3 years after treatment
  Improvement of headache at 3 months, 1 year, and 3 years after treatment Headache was assessed by the WHO pain grading classification:Grade 0: No pain; Grade I: mild pain, intermittent pain, no medication; Grade II: moderate pain, continuous pain, affecting rest, need analgesics; level III: severe pain, continuous pain, need analgesics relieve pain; Grade IV: severe pain, continuous severe pain with changes in blood pressure and pulse.
Improvement of neurological dysfunction | 3 months, 1 year, and 3 years after treatment
  The modified Rankin score was used to evaluate neurological dysfunction: Grade 0, completely asymptomatic; Grade 1, able to complete all daily duties and activities despite symptoms, but without obvious dysfunction; Grade 2, mildly disabled, unable to complete all activities before illness, but does not need help, can take care of themself; Grade 3, moderately disabled, requires some help, but does not need help while walking; Grade 4, severely disabled, unable to walk independently, unable to meet their own needs without help from others; Grade 5, severely disabled, bedridden, incontinence, requiring continuous care And attention; Grade 6, death.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Shuo, MD, Study Chair — Beijing Tiantan Hospital; Li Youxiang, MD, Principal Investigator — Beijing Neurosurgical Institute; Liu Ali, MD, Principal Investigator — Beijing Neurosurgical Institute; Zhao Yuanli, MD, Principal Investigator — Beijing Neurosurgical Institute; Chen Xiaolin, MD, Principal Investigator — Beijing Neurosurgical Institute
Locations (1):
- Capital medical university affiliated Beijing Tiantan hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Meng X, Gao D, He H, Sun S, Liu A, Jin H, Li Y. A Machine Learning Model Predicts the Outcome of SRS for Residual Arteriovenous Malformations after Partial Embolization: A Real-World Clinical Obstacle. World Neurosurg. 2022 Jul;163:e73-e82. doi: 10.1016/j.wneu.2022.03.007. Epub 2022 Mar 9. PMID 35276397
- [Result] Meng X, Gao D, Jin H, Wang K, Bao E, Liu A, Li Y, Sun S. Factors Affecting Volume Reduction Velocity for Arteriovenous Malformations After Treatment With Dose-Stage Stereotactic Radiosurgery. Front Oncol. 2021 Dec 20;11:769533. doi: 10.3389/fonc.2021.769533. eCollection 2021. PMID 34988014
- [Result] Li Z, Chen Y, Chen P, Li R, Ma L, Yan D, Zhang H, Han H, Zhao Y, Zhang Y, Meng X, Jin H, Li Y, Chen X, Zhao Y. Quantitative evaluation of hemodynamics after partial embolization of brain arteriovenous malformations. J Neurointerv Surg. 2022 Nov;14(11):1112-1117. doi: 10.1136/neurintsurg-2021-018187. Epub 2021 Dec 6. PMID 34872987
- [Result] Yan D, Chen Y, Li Z, Zhang H, Li R, Yuan K, Han H, Meng X, Jin H, Gao D, Li Y, Sun S, Liu A, Chen X, Zhao Y. Stereotactic Radiosurgery With vs. Without Prior Embolization for Brain Arteriovenous Malformations: A Propensity Score Matching Analysis. Front Neurol. 2021 Oct 12;12:752164. doi: 10.3389/fneur.2021.752164. eCollection 2021. PMID 34712200
- [Result] Meng X, He H, Liu P, Gao D, Chen Y, Sun S, Liu A, Li Y, Jin H. Radiosurgery-Based AVM Scale Is Proposed for Combined Embolization and Gamma Knife Surgery for Brain Arteriovenous Malformations. Front Neurol. 2021 Mar 30;12:647167. doi: 10.3389/fneur.2021.647167. eCollection 2021. PMID 33859610
- [Result] Chen Y, Meng X, Ma L, Zhao Y, Gu Y, Jin H, Gao D, Li Y, Sun S, Liu A, Zhao Y, Chen X, Wang S. Contemporary management of brain arteriovenous malformations in mainland China: a web-based nationwide questionnaire survey. Chin Neurosurg J. 2020 Sep 1;6:26. doi: 10.1186/s41016-020-00206-0. eCollection 2020. PMID 32922955
- [Result] Chen Y, Li R, Ma L, Meng X, Yan D, Wang H, Ye X, Jin H, Li Y, Gao D, Sun S, Liu A, Wang S, Chen X, Zhao Y. Long-term outcomes of brainstem arteriovenous malformations after different management modalities: a single-centre experience. Stroke Vasc Neurol. 2021 Mar;6(1):65-73. doi: 10.1136/svn-2020-000407. Epub 2020 Sep 14. PMID 32928999
- [Result] Chen Y, Yan D, Li Z, Ma L, Zhao Y, Wang H, Ye X, Meng X, Jin H, Li Y, Gao D, Sun S, Liu A, Wang S, Chen X, Zhao Y. Long-Term Outcomes of Elderly Brain Arteriovenous Malformations After Different Management Modalities: A Multicenter Retrospective Study. Front Aging Neurosci. 2021 Feb 18;13:609588. doi: 10.3389/fnagi.2021.609588. eCollection 2021. PMID 33679374
- [Result] Deng Z, Chen Y, Ma L, Li R, Wang S, Zhang D, Zhao Y, Zhao J. Long-term outcomes and prognostic predictors of 111 pediatric hemorrhagic cerebral arteriovenous malformations after microsurgical resection: a single-center experience. Neurosurg Rev. 2021 Apr;44(2):915-923. doi: 10.1007/s10143-019-01210-4. Epub 2020 Feb 20. PMID 32078085
- [Result] Chen Y, Li R, Ma L, Zhao Y, Yu T, Wang H, Ye X, Wang R, Chen X, Zhao Y. Single-Stage Combined Embolization and Resection for Spetzler-Martin Grade III/IV/V Arteriovenous Malformations: A Single-Center Experience and Literature Review. Front Neurol. 2020 Oct 29;11:570198. doi: 10.3389/fneur.2020.570198. eCollection 2020. PMID 33193013
- [Derived] Yu T, Han H, Ma L, Zhao Y, Zhang Y, Li Y, Wang S, Chen Y, Chen X. Learning curve and embolisation strategy in single-stage surgery combined embolisation and microsurgery for brain arteriovenous malformations: results from a nationwide multicentre prospective registry study. Stroke Vasc Neurol. 2025 Dec 23;10(6):691-701. doi: 10.1136/svn-2025-004051. PMID 40194846
- [Derived] Han H, Gao D, Ma L, Li R, Li Z, Zhang H, Yuan K, Wang K, Zhang Y, Zhao Y, Jin W, Jin H, Meng X, Yan D, Li R, Lin F, Hao Q, Wang H, Ye X, Kang S, Pu J, Shi Z, Chao X, Lin Z, Lu J, Li Y, Zhao Y, Sun S, Chen Y, Chen X, Wang S; Registry of Multimodality Treatment for Brain Arteriovenous Malformation in Mainland China (MATCH). Long-term outcomes of microsurgery and stereotactic radiosurgery as the first-line treatment for arteriovenous malformations: a propensity score-matched analysis using nationwide multicenter prospective registry data. Int J Surg. 2023 Dec 1;109(12):3983-3992. doi: 10.1097/JS9.0000000000000751. PMID 37720924
- [Derived] Li R, Chen P, Han H, Li Z, Chen X, Chen Y, Zhao Y. Association of nidus size and rupture in brain arteriovenous malformations: Insight from angioarchitecture and hemodynamics. Neurosurg Rev. 2023 Aug 31;46(1):216. doi: 10.1007/s10143-023-02113-1. PMID 37650957
- [Derived] Chen Y, Han H, Jin H, Meng X, Ma L, Li R, Li Z, Yan D, Zhang H, Yuan K, Wang K, Zhao Y, Zhang Y, Jin W, Li R, Lin F, Hao Q, Wang H, Ye X, Kang S, Gao D, Pu J, Shi Z, Chao X, Lin Z, Lu J, Li J, Sun S, Liu A, Chen X, Li Y, Zhao Y, Wang S; Registry of Multimodality Treatment for Brain Arteriovenous Malformation in Mainland China (MATCH). Association of embolization with long-term outcomes in brain arteriovenous malformations: a propensity score-matched analysis using nationwide multicenter prospective registry data. Int J Surg. 2023 Jul 1;109(7):1900-1909. doi: 10.1097/JS9.0000000000000341. PMID 37226884
- [Derived] Chen Y, Han H, Ma L, Li R, Li Z, Yan D, Zhang H, Yuan K, Wang K, Zhao Y, Zhang Y, Jin W, Li R, Lin F, Meng X, Hao Q, Wang H, Ye X, Kang S, Jin H, Li Y, Gao D, Sun S, Liu A, Wang S, Chen X, Zhao Y. Multimodality treatment for brain arteriovenous malformation in Mainland China: design, rationale, and baseline patient characteristics of a nationwide multicenter prospective registry. Chin Neurosurg J. 2022 Oct 17;8(1):33. doi: 10.1186/s41016-022-00296-y. PMID 36253875
- [Derived] Li N, Yan D, Li Z, Chen Y, Ma L, Li R, Han H, Meng X, Jin H, Zhao Y, Chen X, Wang H, Zhao Y. Long-term outcomes of Spetzler-Martin grade IV and V arteriovenous malformations: a single-center experience. Neurosurg Focus. 2022 Jul;53(1):E12. doi: 10.3171/2022.4.FOCUS21648. PMID 35901717